CLINICAL TRIAL: NCT03750812
Title: The Effect of Age, Physical Fitness and a Single Bout of Aerobic Exercise on Motor and Cognitive Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0065-18
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity; Age-related Cognitive Decline
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Highly fit older adults - Exercise (Active Comparator): This will receive an aerobic exercise intervention
  Interventions: Behavioral: Aerobic Exercise
- Poorly fit older adults - Exercise (Active Comparator): This arm will receive an aerobic exercise intervention
  Interventions: Behavioral: Aerobic Exercise
- Highly fit young adults - Exercise (Active Comparator): This arm will receive an aerobic exercise intervention
  Interventions: Behavioral: Aerobic Exercise
- Poorly fit young adults - Exercise (Active Comparator): This arm will receive an aerobic exercise intervention
  Interventions: Behavioral: Aerobic Exercise
- Highly fit older adults - TV (Active Comparator): This arm will sit at rest and watch television
  Interventions: Behavioral: Watching television
- Poorly fit older adults - TV (Active Comparator): This arm will sit at rest and watch television
  Interventions: Behavioral: Watching television
- Highly fit young adults - TV (Active Comparator): This arm will sit at rest and watch television
  Interventions: Behavioral: Watching television
- Poorly fit young adults - TV (Active Comparator): This arm will sit at rest and watch television
  Interventions: Behavioral: Watching television

INTERVENTIONS:
Behavioral: Aerobic Exercise — Medium-intense 60% heart rate reserve (HRR) aerobic exercise on a treadmill for 30 minutes
  Arms: Highly fit older adults - Exercise; Highly fit young adults - Exercise; Poorly fit older adults - Exercise; Poorly fit young adults - Exercise
Behavioral: Watching television — Sitting and watching television for 30 minutes
  Arms: Highly fit older adults - TV; Highly fit young adults - TV; Poorly fit older adults - TV; Poorly fit young adults - TV

SUMMARY:
The proposed study is intended to examine the connection between two types of inhibition - cognitive and motor and the connection between motor inhibitory functions and a single bout of physical exercise in the context of age and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Do not take psychiatric drugs on a regular basis
* Geriatric Depression Scale score less than 3
* Mini-Mental State Examination score higher than 27
* Healthy and able to exercise at medium intensity

Exclusion Criteria:

* All others

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in cognitive functions after exercise | One and a half hours
  This improvement will be measured through use of a vocal stroop test
Improvement in motor functions after exercise | One and a half hours
  This improvement will be measured through use of a multi-limb reaction time test

CONTACTS AND LOCATIONS:
Overall Officials: Yael Netz, PhD, Study Director — Wingate Academic Institute
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No